CLINICAL TRIAL: NCT05801393
Title: Combined HRC, CT Cisternography and MR Cisternography in Assessment of Active CSF Rhinorrhes Compared to Operative Findings
Brief Title: HRCT, CT Cisternography and MR Cisternography in Assessment of CSF Rhinorrhea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Abdelsabour Mohamed, GAMohamed, Assiut University
Other Study IDs: cisternography CSF rhinorrhea
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Imaging of Active CSF Rhinorrhea
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CT, MRI — HRCT with no IV contrast administration and bone algorithm. Intra thecal injection of contrast, then CT in prone position to obtain direct coronal cuts.
  MR cisternography using a three dimensional constructive interference in steady state (3D-CISS) sequence.

SUMMARY:
To assess the diagnostic accuracy of combined high resolution CT, CT cisternography and MR cisternography in pre operative assessment of active CSF leak, compared by endoscopic sinus surgery.

DETAILED DESCRIPTION:
CSF rhinorrhea is defined as passage of CSF from the subarachnoid space through osseous and dural defect at skull base into the nasal cavity.

Causes of CSF rhinorrhea are classified into traumatic (including iatrogenic) and non traumatic (including spontaneous leak).

Patients are presented by variable symptoms including clear nasal discharge, headache or with complications like meningitis or even brain abscess, so closure of the defect is of great importance with required accurate localization of the defect and its dimensions.

CSF rhinorrhea can be also classified into active when with active dripping or inactive when dripping is intermittent.

Different imaging modalities have been employed to localize and characterize skull base defects responsible for CSF leakage including computed tomography (CT), CT cisternography (CTC), magnetic resonance imaging (MRI), MR cisternography (MRC) and radionuclide cisternography (RNC). However, there is still no gold standard imaging modality.

High resolution computed tomography (HRCT) provides accurate bone details, but difficult to differentiate para nasal sinus secretions from CSF leak. contrast enhancing CT cisternography has an advantage of definite proof of CSF leak and definite anatomical localization of the bony defect, but side effects like headache and meningeal irritation may occur.

Magnetic resonance imaging (MRI) with 3D- constructive interference in steady state (3D-CISS) (MR cisternography) instead of the invasive CT cisternography shows CSF as a bright signal without intra thecal contrast injection. Also MRI provides intra cranial details, but it lacks of bony details.

In the present prospective study, we will assess the use of HRCT, CTC and MRC imaging modalities in definite diagnosis and localization of active CSF leak.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with active traumatic or non traumatic CSF leakage.
* (2) patients with adequate organ function.

Exclusion Criteria:

* (1) Patients known to have contrast hypersensitivity. (2) Patients with any general contraindication to MRI as presence of para magnetic substance as pacemakers or with claustrophobia.

  (3) Patients with contraindication to lumbar puncture:
  * Infection near the puncture site, fever, sepsis.
  * New focal neurological signs or seizures.
  * Increased intra cranial tension.
  * Space occupying lesion.
  * Vertebral deformity, retropulsion, severe vertebral osteoarthritis or degenerative disc disease renders procedures more technically difficult.
  * Coagulopathy.
  * Patient refusal.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 50 patients with active CSF rhinorrhea, no age limits
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic accuracy of combined high resolution CT, CT cisternography and MR cisternography in pre operative assessment of active CSF leak, compared by endoscopic sinus surgery. | from May 2023 to January 2025
  Patients with persistent or intermittent CSF rhinorrhea will be scanned after a full clinical history with Oto-laryngological examination to confirm the presence of CSF leak